CLINICAL TRIAL: NCT03800537
Title: MR Fingerprinting: A Novel Sequence Applied to Neuroimaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-2071
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2022-08

CONDITIONS: Disease;Neurological
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All Participants (Experimental): All participants will receive the investigational MR Fingerprinting sequence.
  Interventions: Device: MR Fingerprinting

INTERVENTIONS:
Device: MR Fingerprinting — The MR fingerprinting technique requires less than 15 minutes and will be added following the standard MRI sequence.

SUMMARY:
Magnetic Resonance Imaging (MRI) has become one of most important medical imaging tools over the past 30 years because it is non-invasive, requires no ionizing radiation, and provides exquisite images of soft tissues and anatomic structures with many tissue/disease specific contrasts. While MRI has served the community well for many years, it is increasingly clear that it also has significant limitations.

One of the principle limitations is the lack of quantitative information for tissue/structure characterization. The current paradigm of MRI is to use a set of scanner settings to generate an image "weighted" by a specific MR contrast mechanism (physical parameter), where it is hoped that variations in the parameter will be accentuated. However, without quantitative knowledge of the parameters, the final image contrast may depend on many factors, which complicates image interpretation and diagnostic performance. Quantitative measurement can provide a great deal of information about tissue properties and pathological conditions, since these parameters ultimately determine the contrast that is observed in conventional images.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate novel quantitative MRI techniques in clinical studies to determine whether they can provide better, faster and more useful information for clinical diagnosis. Quantitative MRI has been a continuous interest in the MRI community, but extremely challenging due to long acquisition times and sensitivity to motion. Recently, the investigators have introduced a novel MRI data acquisition approach, namely MR Fingerprinting (MRF), for simultaneous measurement of several important parameters in a single MRI scan.

In this study, the investigators propose to apply MR Fingerprinting at UNC and evaluate its performance for different neurological diseases. The investigators hypothesize that the quantitative MR imaging technique will lead to improved tissue characterization and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* The study will include English-speaking patients that are already scheduled to undergo a clinical neurological MRI for diagnostic purposes.

Exclusion Criteria:

* Pregnant women will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Z Lee, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 14
Completed | 10
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Visible Region of Interest (Imaging Visibility)
Description: Magnetic Resonance (MR) fingerprinting sequences will be examined to determine their utility for visualizing pathology.
Time Frame: Immediately following MRI completion, within approximately 5 minutes
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 10
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Throughout the standard of care MRI and including the investigational MRI sequence, a total of up to approximately 25 minutes.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03800537/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT03800537/ICF_001.pdf